CLINICAL TRIAL: NCT04499625
Title: Intraoperative and Postoperative Outcomes of Sinus Floor Elevation Using Lateral Window Technique Versus Hydrodynamic Transalveolar Approach: A Randomized Controlled Trial
Brief Title: Lateral Window Versus Intralift™ Sinus Floor Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B707201316423
Record Dates: First submitted 2020-07-14; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Intraoperative Outcomes; Postoperative Outcomes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Lateral window (Other): Standard surgical technique to access maxillary sinus for sinus floor augmentation procedure.
  Interventions: Procedure: Sinus floor elevation
- Test - Hydrodynamic transalveolar approach (Experimental): Novel transalveolar approach (using an ultrasonic device) to access maxillary sinus for sinus floor augmentation procedure.
  Interventions: Device: Sinus floor elevation using an ultrasonic device

INTERVENTIONS:
Procedure: Sinus floor elevation
  Arms: Control - Lateral window
Device: Sinus floor elevation using an ultrasonic device
  Arms: Test - Hydrodynamic transalveolar approach

SUMMARY:
Several approaches have been used in order to regenerate bone in the upper jaw in case of insufficient alveolar bone height for implant placement. However, new emerging techniques need to be assessed and compared to conventional methods in order to define their potential indications.

The purpose of the present randomized controlled clinical trial was to compare the clinical outcomes of two sinus floor elevation techniques: conventional lateral window technique versus a novel transalveolar approach using hydrodynamic ultrasonic device.

ELIGIBILITY:
Inclusion Criteria:

* edentulism in the posterior maxilla (unitary or plural)
* need of a sinus floor augmentation procedure before implant placement

Exclusion Criteria:

* any uncontrolled systemic disease
* ongoing chemo- or radiotherapy
* history of maxillary sinus diseases or acute sinus-related issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Sinus membrane perforation | During the surgery (from beginning to end)
  Presence/absence of sinus membrane perforation during the surgery
Surgical procedure duration | From beginning of surgery until the end of surgery
  The time measurement started from the administration of local anesthesia and ended when the placement of final suture was completed. The time was measured using a stopwatch.
Edema | From the end of surgery up to 1 week postoperatively
  Presence/absence of edema postoperatively
Hematoma | From the end of surgery up to 1 week postoperatively
  Presence/absence of hematoma postoperatively
Postsurgical bleeding | From the end of surgery up to 1 week postoperatively
  Presence/absence of bleeding postoperatively
Nasal discharge | From the end of surgery up to 1 week postoperatively
  Presence/absence of nasal discharge postoperatively
NSAID consumption | From the end of surgery up to 1 week postoperatively
  Quantification of NSAID consumption per day up to 1 week postoperatively (tablets/per day)
Patient related outcome measures (PROMs) | From right before the surgery up to 1 week postoperatively
  PROMs were assessed with a questionnaire using a visual analogue scale (VAS), which was given to all participants in order to assess their perception before, during, and after the intervention. A graduated scale from 0 to 10 was used, with a lower score presenting a better outcome.

SECONDARY OUTCOMES:
Radiographic outcomes | From the baseline (surgery procedure) up to 1 year post-surgery
  Radiographic (CBCT) qualitative assessment of the gained volume (change in volume from baseline to 1 year postoperatively).
Implant survival rates | From the baseline (surgery procedure) up to 1 year post-surgery
  Implant survival rates assessment at 1 year postoperatively.

REFERENCES:
- [Derived] Bacevic M, Compeyron Y, Lecloux G, Rompen E, Lambert F. Intraoperative and postoperative outcomes of sinus floor elevation using the lateral window technique versus the hydrodynamic transalveolar approach: a preliminary randomized controlled trial. Clin Oral Investig. 2021 Sep;25(9):5391-5401. doi: 10.1007/s00784-021-03847-2. Epub 2021 Mar 10. PMID 33694027